CLINICAL TRIAL: NCT07281794
Title: Clinical Validity of the DANU Sports System for Gait and Balance Assessment in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: DANU Sports Ltd (Unknown)
Responsible Party: Principal Investigator, GabriellaGatti, Postgraduate Research Student, Northumbria University
Other Study IDs: 8543b
Record Dates: First submitted 2025-09-16; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease (PD); Healthy (Controls)
Keywords: DANU; Clinical Validation; Wearable Electronic Devices
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease (PD): Participants with a clinical diagnosis of Parkinson's Disease meeting the described eligibility criteria will be recruited to take part within this study. The aim is to recruit 60 people with Parkinson's.
- Healthy Control (HC): Aged-matched (over 50 years old) healthy controls who meet the described eligibility criteria will be recruited to participate in this study. The aim is to recruit 60 participants.

SUMMARY:
This observational study aims to explore the use of the DANU Smart Socks for gait and balance assessment in people with Parkinson's (PwP). The study will compare walking and balance outcomes produced by DANU from people with Parkinson's (PwP) and a group of healthy individuals of similar age. The project aims to investigate if the gait and balance data collected are linked to measures of Parkinson's symptoms such as disease progression and cognitive abilities. Gait and balance outcomes will be obtained through one observational laboratory visit.

DETAILED DESCRIPTION:
Methods:

Institutional ethics have been obtained (Project ID: 8543). Utilising an observational design, participants will be asked to attend one visit to Northumbria University, Newcastle Upon Tyne.

Visit 1: Participants will complete a series of clinical and cognitive measures including the Movement Disorders Society's-Unified Parkinson's Disease Rating Scale, Montreal Cognitive Assessment, Freezing of Gait Questionnaire and Falls Efficacy Scale to act as descriptive measures. Following this, the investigators will conduct a concurrent data collection throughout a battery of motor tasks. The DANU system will be used alongside APDM Mobility Lab throughout the full duration of data collection. Mobility assessments include a 2-Minute Walk Test, 3 walkway trials, a Timed Up and Go and a series of 2-Minute Balance tasks.

ELIGIBILITY:
Parkinson's Group Inclusion Criteria:- Clinical diagnosis of Parkinson's by a movement disorder specialist according to UK brain bank criteria.

* PD stages I-III (Hoehn and Yahr Rating Scale)
* Able to attend Northumbria University, Newcastle Upon Tyne for study visits.
* Able to walk and stand unassisted for a minimum of 2-minutes.
* Aged 50 years old or over

Parkinson's Group Exclusion Criteria:

* History of neurological disorders other than PD (e.g., Huntington's disease, stroke, traumatic brain injury, multiple sclerosis, Alzheimer's disease etc.)
* Unable to walk or stand unaided.
* Montreal Cognitive Assessment (MoCA) score < 21
* Significant issues unrelated to PD that may affect gait (e.g., musculoskeletal issues, back pain, recent surgery etc.)

Healthy Control Inclusion Criteria:

* Ability to attend Northumbria University, Newcastle Upon Tyne for study visits.
* Aged 50 years old or over.
* Able to walk and stand unassisted for a minimum of 2-minutes.

Healthy Control Exclusion Criteria:

* History of neurological disorders (e.g. Huntington's disease, stroke, traumatic brain injury, multiple sclerosis, Alzheimer's disease etc.)
* Significant issues that may affect walking (e.g., musculoskeletal issues, back pain, recent surgery etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited if they fulfill the exclaimed participation criteria and are located within the North East of England. Participants will be recruited from our existing laboratory database, word of mouth and through visiting local groups.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Stride Length | Outcomes will be obtained in one visit (Day 1).
  (m, mean ± standard deviation)
Step Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation)
Stride Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation)
Cadence | Outcomes will be obtained in one visit (Day 1).
  (steps per minute, mean ± standard deviation)
Ground Contact Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation)
Swing Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation)
Stride Velocity | Outcomes will be obtained in one visit (Day 1).
  (m/s, mean ± standard deviation)
Gait Velocity | Outcomes will be obtained in one visit (Day 1).
  (m/s, mean ± standard deviation)
Area of Ellipse | Outcomes will be obtained in one visit (Day 1).
  (mm², mean ± standard deviation)
Length of Ellipse | Outcomes will be obtained in one visit (Day 1).
  (mm, mean ± standard deviation)
Width of Ellipse | Outcomes will be obtained in one visit (Day 1).
  (mm, mean ± standard deviation)
Total Displacement | Outcomes will be obtained in one visit (Day 1).
  (mm, mean ± standard deviation)
Medio-Lateral Range | Outcomes will be obtained in one visit (Day 1).
  (mm, mean ± standard deviation)
Anterior-Posterior Range | Outcomes will be obtained in one visit (Day 1).
  (mm, mean ± standard deviation)

OTHER OUTCOMES:
Double Support Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation)
Single Support Time | Outcomes will be obtained in one visit (Day 1).
  (s, mean ± standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Vitorio, PhD, Principal Investigator — Northumbria University
Locations (2):
- United Kingdom (2):
  - Northumbria University, Newcastle upon Tyne, Tyne and Wear
  - Northumbria University, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DANU Medical Website: Study Collaborator and Smart Sock System. — https://www.danumedical.com/